CLINICAL TRIAL: NCT02974101
Title: AdaptiveStim Objectifying Subjective Pain Questionnaires
Acronym: EMINENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Moens Maarten, Prof. dr., Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMINENT1
Record Dates: First submitted 2016-11-22; First posted 2016-11-28 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Spinal cord stimulation; AdaptiveStim
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- spinal cord stimulation(RestoreSensor) (Experimental)
  Interventions: Other: registration of AdaptiveStim

INTERVENTIONS:
Other: registration of AdaptiveStim

SUMMARY:
This is a prospective, multi-center, correlation study in which the investigators aim to explore the relationship between subjective pain questionnaires and the AdaptiveStim accelerometer output.

DETAILED DESCRIPTION:
The aim of this research is to gather the necessary information relating to the patient his subjective self-report and the more objective information from the implanted IPG (RestoreSensor). Such subjective information can be gathered from the AdaptivStim output.

The main focus of this study is to explore the relationship between the subjective reporting of functional disability with the ODI, sleep quality with the Actiwatch and PSQI, pain intensity with the NRS-diary and the objective measurement of functional positions with the AdaptiveStim in patients receiving high density spinal cord stimulation.

ELIGIBILITY:
Inclusion Criteria:

* FBSS patients treated with SCS (IPG = RestoreSensor) who achieved a steady state (steady state is considered when the parameters didn't changed for at least one month)
* Age > 18 years

Exclusion Criteria:

* Patients with Parkinson's disease
* Patients immobilised due to limb/pelvis/costal fractures
* Stroke patients with MRS>3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
AdaptiveStim output | The change between baseline (T1) and the second assessment 7 days later (T1+7days)
  The Implantable Pulse Generator contains a processor and accelerometer to record objective information about 7 functional positions.
Disability | Disability will be measured at the second assessment namely 7 days after the first assessment
  Disability will be measured using the Oswestry Disability Index (ODI) questionnaire

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) pain diary | Three times every day (morning, afternoon and evening), during 7 days (from baseline assessment (T1) to second assessment (T1+7days))
Objective sleep quality will be measured using the Actiwatch spectrum plus (Respironics). | Three times every day (morning, afternoon and evening), during 7 days (from baseline assessment (T1) to second assessment (T1+7days))
  This compact and lightweight electronic device similar in size to a wristwatch is worn on the non-dominant hand, and measures and records sleep quality
Subjective sleep quality | Disability will be measured at the second assessment namely 7 days after the first assessment
  Subjective sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI).

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Brussel, Brussels, Vlaams Brabant